CLINICAL TRIAL: NCT00022035
Title: Influenza Vaccine Immunogenicity in Children During and After Therapy for Acute Lymphoblastic Leukemia
Brief Title: Vaccine Therapy in Preventing Flu in Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: RP 99-12; RPCI-RP-9912; NCI-G01-1990
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Infection; Leukemia
Keywords: childhood acute lymphoblastic leukemia in remission; infection
MeSH Terms: conditions — Infections; Leukemia | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: trivalent influenza vaccine

SUMMARY:
RATIONALE: Flu vaccine may help the body build an immune response and decrease the occurrence of flu in children who are receiving chemotherapy for acute lymphoblastic leukemia.

PURPOSE: Clinical trial to study the effectiveness of vaccine therapy in preventing flu in children who have acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the immune response, in terms of the formation of protective antibody titers to influenza, in children with acute lymphoblastic leukemia treated with split-virus trivalent influenza vaccine.
* Correlate the formation of protective antibody titers following immunization with the absolute neutrophil counts and absolute lymphocyte counts in these patients at the time of vaccination.

OUTLINE: This is a multicenter study. Patients are stratified according to current treatment for acute lymphoblastic leukemia (consolidation chemotherapy vs maintenance chemotherapy vs off therapy for the past 6 months).

Patients receive split-virus trivalent influenza vaccine intramuscularly once or twice at 4 weeks apart for 2 doses.

Patients are followed at week 5. Patients receiving 2 doses of vaccine are also followed at week 9.

PROJECTED ACCRUAL: A total of 175 patients (50 receiving consolidation therapy, 75 receiving maintenance therapy, and 50 off therapy) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia

  * In first remission after completion of induction chemotherapy
  * Currently on active treatment OR
  * Completed treatment within the past 6 months

PATIENT CHARACTERISTICS:

Age:

* 1 to 20 at time of diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Pulmonary:

* No acute respiratory distress

Other:

* No history of Guillain-Barre syndrome
* No history of hypersensitivity to chicken eggs, egg products, or components of influenza virus vaccine, including thimerosal
* No febrile illness with fever over 100.4 degrees F
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 7 days since prior antibiotic or antiviral therapy except prophylactic antibiotics

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-08; Primary Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin L. Brecher, MD, Study Chair — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York